CLINICAL TRIAL: NCT04515277
Title: Double-blind, Randomized, Controlled, Three-way Cross-over Study to Evaluate the Effect of Gum Acacia (FibregumTM) on Post-prandial Glucose and Insulin Levels and Food Intake
Brief Title: Study to Evaluate the Effect of Gum Acacia (FibregumTM) on Post-prandial Glucose, Insulin Levels and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nexira (Industry)
Collaborators: Analyze & Realize (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEX/005519
Record Dates: First submitted 2020-08-07; First posted 2020-08-17 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Healthy; Overweight
Keywords: gum acacia; post-prandial glucose (PPG); post-prandial insulin (PPI); blood glucose incremental; appetite sensation; E 414; food additive; FibregumTM; appetite; dietary fibre
MeSH Terms: conditions — Overweight | interventions — Gum Arabic

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, controlled, three-way cross-over design, monocentric nutritional study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 40 g (D1) (Active Comparator): 40 g gum acacia powder (D1). Treatment type is applied with the standardized breakfast (in 300 mL orange juice) on the test days (V2, V3 or V4).
  Interventions: Dietary Supplement: 40 g Gum acacia (FibregumTM)
- 20 g (D2) (Active Comparator): 20 g gum acacia powder (D2). Treatment type is applied with the standardized breakfast (in 300 mL orange juice) on the test days (V2, V3 or V4).
  Interventions: Dietary Supplement: 20 g Gum acacia (FibregumTM)
- No treatment (NT) (Other): 0 g gum acacia powder. Standardized breakfast (in 300 mL orange juice) on the test days (V2, V3 or V4).
  Interventions: Dietary Supplement: 0 g Gum acacia (FibregumTM)

INTERVENTIONS:
Dietary Supplement: 40 g Gum acacia (FibregumTM) — Applied in 300 mL of orange juice with breakfast (single use at visit)
  Other Names: D1
  Arms: 40 g (D1)
Dietary Supplement: 20 g Gum acacia (FibregumTM) — Applied in 300 mL of orange juice with breakfast (single use at visit)
  Other Names: D2
  Arms: 20 g (D2)
Dietary Supplement: 0 g Gum acacia (FibregumTM) — 300 mL of orange juice with breakfast (single use at visit)
  Other Names: no treatment
  Arms: No treatment (NT)

SUMMARY:
Study to evaluate the effect of gum acacia (FibregumTM) on post-prandial glucose and insulin levels and food intake in normal-weight and overweight subjects during a 2-7 weeks intervention period. In addition, tolerability and safety of gum acacia (FibregumTM) will be assessed.

DETAILED DESCRIPTION:
Gum arabic is a heteropolysaccharide (molecular weight 350-850 kDa) harvested from Acacia seyal or Acacia senegal. It is highly soluble and broadly used in numerous solid and liquid food matrices.

For the assessment of non-digestible carbohydrates as dietary fiber, it is eminent to demonstrate that its consumption is related to a specific beneficial physiological effect shown in an appropriate clinical study. The aim of the present trial was to expand the clinical evidence with respect to beneficial effects of gum acacia on post-prandial blood glucose levels, post-prandial insulin levels and prospective ad libitum food intake, in normal-weight and overweight subjects.

The present double-blind, randomized, controlled, three-way cross-over study was to evaluate the effect of gum acacia versus no treatment on post-prandial glucose (PPG) levels in normal-weight and overweight subjects during a 2-7 weeks intervention period.

Additionally, post-prandial insulin (PPI) levels, prospective ad libitum food intake, as well as the safety and tolerability of gum acacia were assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women from 25 to 60 years old
2. Body mass index (BMI) 18.5 kg/m2 - 29.9 kg/m2
3. Generally in good health
4. Normal fasting blood glucose (FBG) 3.9 to <5.6 mmol/L (70 to <100 mg/dL) and HbA1c of 4 to <5.7 %
5. Regularly consuming 3 main meals/day, with breakfast and lunch as dominant meals
6. Familiar with components of the study meals, no disliking and/or extreme preferences for any of the items
7. Readiness to comply with study procedures, in particular:

   * adhere to the defined restrictions prior to / procedures on the test days
   * maintain the habitual level of physical activity and sleep habits during the study
   * fill out the study diary
8. Stable body weight in the last 3 months prior to V1 (≤3% self-reported change)
9. Stable concomitant medications (if any) for at least last 3 months prior to V1
10. Women of childbearing potential:

    * commitment to use contraception methods
    * negative pregnancy testing (beta human chorionic gonadotropin test in urine) at V1
11. Readiness not to participate in another clinical study during this study

Exclusion Criteria:

1. Known allergy or hypersensitivity to the components of the investigational product / study meals
2. History and/or presence of clinically significant self-reported disorder as per investigator's judgement:

   * untreated or non-stabilized thyroid gland disorder
   * untreated or non-stabilized hypertension (regular systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg)
   * digestion/absorption disorders of the gastrointestinal tract (e.g. inflammatory bowel disease, coeliac disease, pancreatitis etc.) and/or GI surgery
   * diabetes mellitus
   * sleep disorder
   * acute or chronic psychiatric disorder
   * any other organ or systemic diseases that could influence the conduct and/or outcome of the study and/or could affect the tolerability of the subject
3. Subjects with difficult vein access or sensitive to blood draws
4. Nighttime eating/snacking (after 10 pm)
5. Excessive consumption of artificial sweeteners (e.g. in beverages)
6. History and/or presence of eating disorders like bulimia, anorexia nervosa, binge-eating as per investigator's judgement
7. Use of treatment/supplementation in the last 2 months prior to V1 and during the study, as per investigator's judgment, that could influence gastrointestinal functions, body weight, blood glucose levels or otherwise interfere with study conduct / evaluation
8. Deviation of safety laboratory parameter(s) at V1 (except for Hb and HbA1c) that is:

   * clinically significant or
   * >2x upper limit of normal, unless the deviation is justified by a previously known not clinically relevant condition (e.g. Gilbert's syndrome)
9. Diet/weight loss programs within the last 3 months prior to V1 and during the study
10. Recent blood donation within the last 1 month prior to study
11. Smoking within the last 6 months prior to V1 and during the study
12. Vegetarian, vegan or other restrictive diet
13. Night shift work
14. History or current abuse of alcohol, drug and/or medication
15. Women of child-bearing potential: pregnancy or nursing
16. Inability to comply with study procedures
17. Participation in another study during the last 30 days prior to V1
18. Any other reason deemed suitable for exclusion, per investigator's judgment

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Difference in blood glucose incremental AUC 0-120 min between D1 verum group and no treatment group | 2 -7 weeks
  Venous blood samples were drawn for the determination of glucose values, with sampling times at -15 min and immediately prior to the intake of the standardized breakfast (time "0") as well as 15, 30, 45, 60, 90 and 120 min after the "0 min" blood draw.

SECONDARY OUTCOMES:
Difference in blood glucose incremental AUC 0-120 min between D2 verum group and no treatment group | 2 -7 weeks
  Venous blood samples were drawn for the determination of glucose values, with sampling times at -15 min and immediately prior to the intake of the standardized breakfast (time "0") as well as 15, 30, 45, 60, 90 and 120 min after the "0 min" blood draw.
Food (energy) intake at ad libitum lunch, in comparison between each verum group vs no treatment group | 2 -7 weeks
  Food was weighed before the subject consumed the meal and afterwards and the energy content of the food consumed was determined.
Individual appetite sensation items (VAS for satiety, hunger, fullness, prospective consumption, desire to eat), in comparison between each verum group vs no treatment group - VAS values at all time points 0, 15, 30, 45, 60, 90, 120, 180, 210, 240 min | 2 -7 weeks
  Visual analogue scales (VAS) for satiety, hunger, fullness, prospective consumption, desire to eat will be reported as follows:
  Subjects had to record their appetite sensation before and after consumption of the standardised breakfast provided on site. VAS, 100-mm in length, were used to assess the following items:
  * Hunger: How hungry are you? (Not at all <-> Extremely / As hungry as I have ever felt)
  * Fullness: How full are you? (Not at all <-> Extremely / As full as I have ever felt)
  * Satiety: How satiated are you? (Not at all <-> Extremely)
  * Desire to eat (appetite): How strong is your desire to eat? (Very weak / Extremely low <-> Very strong / Extremely high)
  * Prospective consumption (Quantity): How much do you think you could (or would want to) eat right now? (Nothing at all <-> A very large amount)
Individual appetite sensation items (VAS for satiety, hunger, fullness, prospective consumption, desire to eat), in comparison between each verum group vs no treatment group - maximal/minimal VAS values | 2 -7 weeks
  Visual analogue scales (VAS) for satiety, hunger, fullness, prospective consumption, desire to eat will be reported as follows:
  Subjects had to record their appetite sensation before and after consumption of the standardised breakfast provided on site. VAS, 100-mm in length, were used to assess the following items:
  * Hunger: How hungry are you? (Not at all <-> Extremely / As hungry as I have ever felt)
  * Fullness: How full are you? (Not at all <-> Extremely / As full as I have ever felt)
  * Satiety: How satiated are you? (Not at all <-> Extremely)
  * Desire to eat (appetite): How strong is your desire to eat? (Very weak / Extremely low <-> Very strong / Extremely high)
  * Prospective consumption (Quantity): How much do you think you could (or would want to) eat right now? (Nothing at all <-> A very large amount)
Individual appetite sensation items (VAS for satiety, hunger, fullness, prospective consumption, desire to eat), in comparison between each verum group vs no treatment group - total AUC 0-15, 0-30, 0-45, 0-60, 0-90, 0-120, 0-180, 0-210, 0-240 min | 2 -7 weeks
  Visual analogue scales (VAS) for satiety, hunger, fullness, prospective consumption, desire to eat will be reported as follows:
  Subjects had to record their appetite sensation before and after consumption of the standardised breakfast provided on site. VAS, 100-mm in length, were used to assess the following items:
  * Hunger: How hungry are you? (Not at all <-> Extremely / As hungry as I have ever felt)
  * Fullness: How full are you? (Not at all <-> Extremely / As full as I have ever felt)
  * Satiety: How satiated are you? (Not at all <-> Extremely)
  * Desire to eat (appetite): How strong is your desire to eat? (Very weak / Extremely low <-> Very strong / Extremely high)
  * Prospective consumption (Quantity): How much do you think you could (or would want to) eat right now? (Nothing at all <-> A very large amount)
Individual appetite sensation items (VAS for satiety, hunger, fullness, prospective consumption, desire to eat), in comparison between each verum group vs no treatment group - incremental AUC 0-15, 0-30, 0-45, 0-60, 0-90, 0-120, 0-180, 0-210, 0-240 min | 2 -7 weeks
  Visual analogue scales (VAS) for satiety, hunger, fullness, prospective consumption, desire to eat will be reported as follows:
  Subjects had to record their appetite sensation before and after consumption of the standardised breakfast provided on site. VAS, 100-mm in length, were used to assess the following items:
  * Hunger: How hungry are you? (Not at all <-> Extremely / As hungry as I have ever felt)
  * Fullness: How full are you? (Not at all <-> Extremely / As full as I have ever felt)
  * Satiety: How satiated are you? (Not at all <-> Extremely)
  * Desire to eat (appetite): How strong is your desire to eat? (Very weak / Extremely low <-> Very strong / Extremely high)
  * Prospective consumption (Quantity): How much do you think you could (or would want to) eat right now? (Nothing at all <-> A very large amount)
Composite score ([desire to eat + hunger + (100-fullness) + prospective consumption]/4), in comparison between each verum group vs no treatment group - VAS values at all time points 0, 15, 30, 45, 60, 90, 120, 180, 210, 240 min | 2 -7 weeks
  Composite score is calculated as follows:([desire to eat + hunger + (100 - satiety) + estimated consumption]/4).
  Subjects had to record their appetite sensation before and after consumption of the standardised breakfast provided on site. Visual analogue scales (VAS), 100-mm in length, were used to assess the following items:
  * Hunger: How hungry are you? (Not at all <-> Extremely / As hungry as I have ever felt)
  * Satiety: How satiated are you? (Not at all <-> Extremely)
  * Desire to eat (appetite): How strong is your desire to eat? (Very weak / Extremely low <-> Very strong / Extremely high)
  * Prospective consumption (Quantity): How much do you think you could (or would want to) eat right now? (Nothing at all <-> A very large amount)
Composite score ([desire to eat + hunger + (100-fullness) + prospective consumption]/4), in comparison between each verum group vs no treatment group - maximal/minimal VAS values | 2 -7 weeks
  Composite score is calculated as follows:([desire to eat + hunger + (100 - satiety) + estimated consumption]/4).
  Subjects had to record their appetite sensation before and after consumption of the standardised breakfast provided on site. Visual analogue scales (VAS), 100-mm in length, were used to assess the following items:
  * Hunger: How hungry are you? (Not at all <-> Extremely / As hungry as I have ever felt)
  * Satiety: How satiated are you? (Not at all <-> Extremely)
  * Desire to eat (appetite): How strong is your desire to eat? (Very weak / Extremely low <-> Very strong / Extremely high)
  * Prospective consumption (Quantity): How much do you think you could (or would want to) eat right now? (Nothing at all <-> A very large amount)
Composite score ([desire to eat + hunger + (100-fullness) + prospective consumption]/4), in comparison between each verum group vs no treatment group - total AUC 0-15, 0-30, 0-45, 0-60, 0-90, 0-120, 0-180, 0-210, 0-240 min | 2 -7 weeks
  Composite score is calculated as follows:([desire to eat + hunger + (100 - satiety) + estimated consumption]/4).
  Subjects had to record their appetite sensation before and after consumption of the standardised breakfast provided on site. Visual analogue scales (VAS), 100-mm in length, were used to assess the following items:
  * Hunger: How hungry are you? (Not at all <-> Extremely / As hungry as I have ever felt)
  * Satiety: How satiated are you? (Not at all <-> Extremely)
  * Desire to eat (appetite): How strong is your desire to eat? (Very weak / Extremely low <-> Very strong / Extremely high)
  * Prospective consumption (Quantity): How much do you think you could (or would want to) eat right now? (Nothing at all <-> A very large amount)
Composite score ([desire to eat + hunger + (100-fullness) + prospective consumption]/4), in comparison between each verum group vs no treatment group - incremental AUC 0-15, 0-30, 0-45, 0-60, 0-90, 0-120, 0-180, 0-210, 0-240 min | 2 -7 weeks
  Composite score is calculated as follows:([desire to eat + hunger + (100 - satiety) + estimated consumption]/4).
  Subjects had to record their appetite sensation before and after consumption of the standardised breakfast provided on site. Visual analogue scales (VAS), 100-mm in length, were used to assess the following items:
  * Hunger: How hungry are you? (Not at all <-> Extremely / As hungry as I have ever felt)
  * Satiety: How satiated are you? (Not at all <-> Extremely)
  * Desire to eat (appetite): How strong is your desire to eat? (Very weak / Extremely low <-> Very strong / Extremely high)
  * Prospective consumption (Quantity): How much do you think you could (or would want to) eat right now? (Nothing at all <-> A very large amount)
24 hour energy intake on test days: breakfast+ad libitum lunch+diary records, in comparison between each verum group vs no treatment group | 2 -7 weeks
  After each of the site visits on test days, food and beverage intake during the time period until 24 hours after start of site visit had to be documented by the subjects in the study diary and the energy.
PPG, in comparison between each verum group vs no treatment group - concentration at all time points 0, 15, 30, 45, 60, 90, 120, 180 min | 2 -7 weeks
  Venous blood samples were drawn for the determination of glucose values
PPG, in comparison between each verum group vs no treatment group - maximal concentration | 2 -7 weeks
  Venous blood samples were drawn for the determination of glucose values
PPG, in comparison between each verum group vs no treatment group - total AUC 0-15, 0-30, 0-45, 0-60, 0-90, 0-120, 0-180 min | 2 -7 weeks
  Venous blood samples were drawn for the determination of glucose values
PPG, in comparison between each verum group vs no treatment group - incremental AUC 0-15, 0-30, 0-45, 0-60, 0-90, 0-180 min | 2 -7 weeks
  Venous blood samples were drawn for the determination of glucose values
PPI, in comparison between each verum group vs no treatment group - concentration at all time points 0, 15, 30, 45, 60, 90, 120, 180 min | 2 -7 weeks
  Venous blood samples were drawn for the determination of insulin values
PPI, in comparison between each verum group vs no treatment group - maximal concentration | 2 -7 weeks
  Venous blood samples were drawn for the determination of insulin values
PPI, in comparison between each verum group vs no treatment group - total AUC 0-15, 0-30, 0-45, 0-60, 0-90, 0-120, 0-180 min | 2 -7 weeks
  Venous blood samples were drawn for the determination of insulin values
PPI, in comparison between each verum group vs no treatment group - incremental AUC 0-15, 0-30, 0-45, 0-60, 0-90, 0-120, 0-180 min | 2 -7 weeks
  Venous blood samples were drawn for the determination of insulin values
Global evaluation (by 4-point scale) of benefit by subject and the investigator, in comparison between each verum group vs no treatment group | 2 -7 weeks
  The investigators had to evaluate the benefit of the treatment type (global scaled evaluation with "very good", "good", "moderate" and "poor").

OTHER OUTCOMES:
Gastrointestinal tolerability evaluation (by 4-point scale), in comparison between each verum group and no treatment group | 2 -7 weeks
  Gastrointestinal tolerabilty was assessed by assessing the items burping, cramping, distension, flatulence, nausea, vomiting scored by means of a 4-point scale: 1=none, 2=mild, 3=moderate, 4=severe, on test days only, at 0 min (before the standardized breakfast) and at 1, 2, 3, 4, 6, 12 and 24 hours after intake of standardized breakfast in the subject diary
Blood pressure (systolic and diastolic), in comparison between each verum group and no treatment group | 2 -7 weeks
  Sitting blood pressure (systolic and diastolic) was measured using standard procedures
Pulse rate, in comparison between each verum group and no treatment group | 2 -7 weeks
  Sitting pulse rate was measured using standard procedures
Global evaluation (by 4-point scale) of tolerability by subject and investigator at study end, in comparison between each verum group and no treatment group | 2 -7 weeks
  The investigators had to evaluate the tolerability of the treatment type (global scaled evaluation with "very good", "good", "moderate" and "poor").
Assessment of adverse events throughout the study | 2 -7 weeks
  Any adverse event (AE) that occured during the course of the clinical study had to be recorded
Body weight, in comparison between each verum group and no treatment group | 2 -7 weeks
  Body weight (kg) was measured in subjects in fasting condition wearing only underwear and barefoot, after emptying the bladder and bowels as needed, using standardized weighing scales (Tanita BC-420MA).
Changes in dietary habits, physical activities and sleep habits by questioning, in comparison between each verum group and no treatment group | 2 -7 weeks
  The subjects were questioned with respect to any changes:
  * in their dietary habits (e.g lower/higher calorie intake)
  * in their sleep habits (e.g less/more sleep)
  * in their level of physical activity (e.g lower/higher activity level)

CONTACTS AND LOCATIONS:
Locations (1):
- Analyze & Realize, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No